CLINICAL TRIAL: NCT03397342
Title: MRI-only Radiation Therapy Workflow With Continuous Positive Airway Pressure (CPAP) for Motion Management in the Abdomen
Brief Title: MRI Only Radiation Therapy With CPAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated prematurely well short of enrollment target. Only 5 health participants were enrolled
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-7745
Record Dates: First submitted 2017-05-08; First posted 2018-01-12 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma Liver; Carcinoma, Pancreatic
MeSH Terms: conditions — Carcinoma, Hepatocellular; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- standard breath hold (No Intervention): 1. Breath-hold CT and 4D-CT without CPAP
  2. Breath-hold MRI and 4D-MRI without CPAP a) T1-weighted, T2-weighted, Dixon fat/water, and ultra-short TE images
- CPAP intervention (Experimental): 1. Breath-hold CT without CPAP
  2. 4D-CT with and without CPAP
  3. 4D-MRI with CPAP
     1. T1-weighted, T2-weighted, Dixon fat/water, and ultra-short TE images
  Interventions: Device: CPAP machine

INTERVENTIONS:
Device: CPAP machine — Use of CPAP machine during MRI
  Arms: CPAP intervention

SUMMARY:
The goal of this imaging study is to evaluate and improve the treatment planning techniques for abdominal radiation therapy. To accurately treat a tumor with radiation, Computed Tomography (CT) and Magnetic Resonance Images (MRI) are used to distinguish a tumor from normal, healthy tissue. However the quality of these images can be distorted by motion from breathing. To decrease motion, a patient may be asked to hold their breath or compress the abdomen, but currently there is no standard or best management option for all patients.

This study will explore the use continuous positive airway pressure (CPAP), a pressurized breathing mask, during MRI or CT imaging to decrease motion in the abdomen and produce higher quality images. With these additional images, we will also explore the feasibility of creating treatment plans using the CPAP MRI images alone.

DETAILED DESCRIPTION:
Patients will undergo both CT and MRI prior to abdominal radiation therapy and CBCT and orthogonal kV/MV images prior to each treatment delivery. A two arm study will be performed and patients will be enrolled into a given arm according to their eligibility. Arm 1 is for patients that are either not eligible for CPAP or that are unable to tolerate CPAP. These patients will undergo breath-hold and 4D imaging for both CT and MRI without CPAP. Arm 2 is for patients that are eligible for CPAP and able to tolerate CPAP. These patients will undergo breath-hold CT without CPAP, 4D-CT with and without CPAP and 4D-MRI with CPAP. Two specific aims will be investigated. In Aim 1, we will explore the feasibility of using a MRI-only in Radiation Oncology workflow. A probabilistic classification method will be utilized to generate a pseudo-CT from MRI to support treatment planning and image guidance for radiation therapy. The quality of the pseudo-CT will be evaluated by comparing it with CT. In addition, the reverse mapping will be investigated to create pseudo-MRI from CBCT to improve visualization of treatment targets and soft tissue prior to treatment delivery. In Aim 2, we will evaluate the utility of CPAP as a novel motion reduction methodology for patients with liver and pancreas cancer, to this end CT images with and without CPAP will be used. The evaluation will be based on the changes of motion magnitude, the achievable volumetric reduction in treatment target volumes, and doses to the targets and critical organs.

ELIGIBILITY:
Inclusion Criteria:

* Patients have liver or pancreas tumors (either primary tumors or metastases) and are scheduled to be treated with radiotherapy (either 3D conformal or intensity-modulation radiotherapy (IMRT) with conventional or hypo- fractionation).
* KPS > 70
* If a biopsy is performed, the patient is at least 1 week post-biopsy.
* The patient's age must exceed 18 years.
* The patients must be able to commit to T1-weighted, T2-weighted, Dixon fat and water, ultrashort-TE, and other clinical or research MR sequence images prior to treatment.
* CPAP Eligibility: CPAP is a safe, effective form of therapy with rare complications. Relative contraindications include patients with bullous lung disease, fibrotic lung disease, Claustrophobia and recurrent sinus or ear infections. The absolute contraindications include obtundation /unconsciousness, chest wall trauma, suspected pneumothorax, persistent nausea/vomiting, active upper GI bleeding, history of recent gastric surgery, facial anomalies/trauma [15,16]. If there is any question about the above history and medical problems, the subject will be referred to a pulmonologist for consultation.
* The patients with above contraindications are not CPAP eligible and are enrolled in Arm 1 for the protocol without CPAP
* The eligible patients are enrolled in Arm 2 for the protocol with CPAP.

Exclusion Criteria:

* Any medical condition, which would make the imaging studies unsafe or poorly tolerated
* Known allergic reaction to contrast or shellfish
* Implanted metal devices or foreign bodies that serve as a contraindication to MR imaging
* Creatinine > 1.4 mg/dl and Creatinine clearance < 20 mg/dl.
* Uncontrolled, clinically significant cardiac arrhythmias
* Severe claustrophobia
* Pregnant female
* KPS <70

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhur Garg, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five healthy volunteers were enrolled into the study prior to termination
Groups:
- Standard Breath Hold (4D-MRI Without CPAP): 1. Breath-hold CT and 4D-CT without CPAP
  2. Breath-hold MRI and 4D-MRI without CPAP a) T1-weighted, T2-weighted, Dixon fat/water, and ultra-short TE images
- CPAP Intervention (4D-MRI With CPAP): 1. Breath-hold CT without CPAP
  2. 4D-CT with and without CPAP
  3. 4D-MRI with CPAP
     1. T1-weighted, T2-weighted, Dixon fat/water, and ultra-short TE images
  CPAP machine: Use of CPAP machine during MRI
Period: Overall Study
Arm/Group | Standard Breath Hold (4D-MRI Without CPAP) | CPAP Intervention (4D-MRI With CPAP)
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 5 healthy volunteers were enrolled into the 4D-MRI without CPAP arm prior to discontinuation/termination of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Breath Hold (4D-MRI Without CPAP) | CPAP Intervention (4D-MRI With CPAP) | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Customized [Count of Participants; unit: Participants]
  18-29 years old | 5 | 0 | 5
  20-29 years old | 0 | 0 | 0
  30-39 years old | 0 | 0 | 0
  40-49 years old | 0 | 0 | 0
  50+ years old | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  | 4
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 3 |  | 3
  Unknown or Not Reported | 2 |  | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 4 |  | 4
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Internal Target Volume on 4D-MR and 4D-CT
Description: The primary endpoint of aim 1 is that for the subjects enrolled in the study there is no statistically significant difference in ITV (internal target volumes) between subjects whose treatment is planned with MRI compared to subjects whose treatment is planned with 4D-CT.
Time Frame: baseline
Population: Internal target volume (ITV) assessments were not conducted as only healthy volunteers were enrolled into the study. There is no data to report.
Arm/Group | Standard Breath Hold (4D-MRI Without CPAP) | CPAP Intervention (4D-MRI With CPAP)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Reduction of Tumor Motion Using Continuous Positive Airway Pressure
Description: The primary end point of aim 2 is that for the subjects enrolled in Continuous Positive Airway Pressure (CPAP) arm an average tumor motion reduction of at least 12% can be achieved when CPAP is used compared to free breathing.
Time Frame: baseline
Population: No participants were enrolled into the arm/group entailing 4D-MRI with CPAP and, as such, there is no tumor motion data to evaluate.
Arm/Group | Standard Breath Hold (4D-MRI Without CPAP) | CPAP Intervention (4D-MRI With CPAP)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected initiation of MRI scan to discharge from facility, up to 4 hours
Description: 5 healthy volunteers were enrolled into the MRI only (no CPAP) arm/group prior to study termination.
Arm/Group | Standard Breath Hold (4D-MRI Without CPAP) | CPAP Intervention (4D-MRI With CPAP)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 0/5 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT03397342/Prot_SAP_000.pdf